CLINICAL TRIAL: NCT00851422
Title: Accurate Measurement of Cardiac Output Using the Ultrasound Dilution Technique
Acronym: BCM
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-COSTATUS-5A-H; 2R44HL061994-04A2 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Cardiac Output
Keywords: Ultrasound Dilution; Cardiac Output; Validation of measured ultrasound dilution cardiac output

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Accurate cardiac output determination is a commonly used and important index of myocardial performance. The thermodilution method using a pulmonary artery catheter is the most common approach to cardiac output determination; however, placement of the pulmonary artery catheter is not without risk and at times can be problematic. Ultrasound dilution measurement has been shown to correlate with measured cardiac output in animal models and adults, but it has not been validated in pediatric patients. This study will validate the accuracy of ultrasound dilution measurements of cardiac output to thermodilution measurements of cardiac output in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Transplant patients undergoing hemodynamic evaluation in the catheterization laboratory that are less than 18 years of age and have structurally normal hearts.

Exclusion Criteria:

* Patient's age greater than 18 years, and any structural abnormality of the heart.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Any pediatric patient (aged < 18 years) who has undergone cardiac transplantation and is already scheduled for a biopsy will be offered the opportunity to participate.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Validation of cardiac output measured by ultrasound dilution with cardiac output measured by thermodilution. | 5-8 minutes minimum

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery J Kim, MD, Principal Investigator — Texas Children's Hospital, Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416
- [Result] Crittendon I 3rd, Dreyer WJ, Decker JA, Kim JJ. Ultrasound dilution: an accurate means of determining cardiac output in children. Pediatr Crit Care Med. 2012 Jan;13(1):42-6. doi: 10.1097/PCC.0b013e3182196804. PMID 21499176